CLINICAL TRIAL: NCT04229693
Title: Proteomics of Cerebrospinal Fluid of Preterm Infants With Posthemorrhagic Hydrocephalus With Focus on Intranasal Breast Milk.
Brief Title: Cerebrospinal Fluid Proteom in Dependence of Intranasal Breast Milk
Acronym: NAMU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital of Cologne (Other)
Responsible Party: Principal Investigator, Titus Keller, MD, Principal Investigator, University Hospital of Cologne
Other Study IDs: UHC_NAMU
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Hydrocephalus in Infants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cerebrospinal fluid samples which are collected after routine drainage via ventricle reservoir
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention, only observational.

SUMMARY:
Investigation of the cerebrospinal fluid proteom in preterm infants with posthemorrhagic hydrocephalus in our neonatology center with analysis for modulation of proteom in dependence of breastmilk feeding and way of application such as via gavage tube, oral or nasal application.

DETAILED DESCRIPTION:
Since the nasal route might be highly effective for neurotrophins and other growth factors the cerebrospinal fluid will be investigated using mass spectrometry to identify modulating effects of intranasal breast milk application on the cerebrospinal fluid proteom.

ELIGIBILITY:
Inclusion Criteria:

* preterm infant with hydrocephalus and regular drainage

Exclusion Criteria:

* Inborn error of metabolism

Ages: 3 Days to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All preterm infants at our neonatologic center with hydrocephalus in need of drainage are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-02-07 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Cerebrospinal fluid proteom | weeks
  Cerebrospinal fluid analysis using mass spectrometry including proteomic analysis for differences in dependence of intranasal breast milk application

CONTACTS AND LOCATIONS:
Overall Officials: Titus Keller, MD, Principal Investigator — University of Cologne, Children's Hospital
Locations (1):
- Neonatology at the University Hospital of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keller T, Korber F, Oberthuer A, Schafmeyer L, Mehler K, Kuhr K, Kribs A. Intranasal breast milk for premature infants with severe intraventricular hemorrhage-an observation. Eur J Pediatr. 2019 Feb;178(2):199-206. doi: 10.1007/s00431-018-3279-7. Epub 2018 Nov 1. PMID 30386923